CLINICAL TRIAL: NCT00817752
Title: Ashwagandha: Effects on Stress, Inflammation and Immune Cell Activation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Collaborators: Helfgott Research Institute (Unknown)
Responsible Party: Heather Zwickey, PhD., Helfgott Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 02202007A
Record Dates: First submitted 2009-01-02; First posted 2009-01-06 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2009-01

CONDITIONS: Inflammation; Cancer; Autoimmune Diseases
Keywords: stress; inflammation; natural remedy; cytokines; interleukin; inflammatory conditions; auto-immune disorders
MeSH Terms: conditions — Inflammation; Neoplasms; Autoimmune Diseases | interventions — Ashwagandha

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Receives Ashwagandha herb.
  Interventions: Dietary Supplement: Ashwagandha

INTERVENTIONS:
Dietary Supplement: Ashwagandha — Participants consume 3mL of Ashwagandha for 5 days. Blood work/immune cells (CD4 T-cells, CD8 T-cells, B-cells, NK cells, macrophages, IL-1, IL-6 and TNF-alpha) and psychological assessments (POMS and STAI Self-Evaluation) given at specified time intervals.

SUMMARY:
Ayurvedic medicine has been practiced in for more than 2,500 years. Ashwagandha is one of the most widely utilized herbs in the system. It is thought to affect the endocrine, immune, nervous, and cardiopulmonary systems. This study is designed as a preliminary investigation of the effects of Ashwagandha on stress, inflammation, and immune modulation. Participants will take the liquid extract in cow's milk twice a day for five days. The results of initial, one-day, and final blood draws will be compared to determine participant's beginning and ending levels of cortisol, inflammatory cytokines, and immune-cell activation (CD4 T-cells, CD8 T-cells, B cells and natural killer cells). Measurements will be completed using flow cytometry and ELISA assay. The purpose of this study is to determine which effects of Ashwagandha are most suitable for further investigation.

DETAILED DESCRIPTION:
Due to the increased use of alternative medicine, supplements and herbs are consumed more frequently in the treatment of common ailments. This pilot study investigates the immune, anti-inflammatory and anti-stress effects of Ashwagandha in human subjects.

Liquid extract of the herb will be taken followed by milk; this mode of administration will be used as it approximates the traditional administration as well as making self administration easier for participants. Extract will be taken in 3 milliliter quantities 2 times per day, (morning and evening), for five days. Total dosage of 6 milliliters will approximate the higher end of the traditional daily dosage of 6 grams daily of powdered root.

Flow of visit:

25 participants will arrive at the research lab and after being consented, filling out health histories and two stress questionnaires, (POMS and STAI Self-Evaluation), average milk intake questionnaire. The 25 participants will receive blood draws. They will then be administered the herb extract, milk and instructions for taking them.

Subjects will return to the research institute after 24 hours for a second blood draw and then after 5 days for a final blood draw and two more stress questionnaires, (POMS and STAI Self-Evaluation).

Once the blood samples are drawn, they will be refrigerated and processed within 24 hours at the NCNM laboratory. Initially they will be centrifuged to separate the white from the red blood cells using Ficoll separating tubes. Then the white blood cells will be stained using CD69 marker (Cytokine Detection type 69) which assesses cell-surface phenotypic markers in combination with intracellular cytokines, measuring response to activation. It is especially effective for rare-event, antigen-specific events, such as the administration of a specific immune-stimulating herbal tincture. We will also stain with other similar florescent CD markers specific for CD4 T-cells, CD8 T-cells, B-cells, NK cells, and macrophages. These markers will be analyzed using a FACScan flow cytometer, which will count the number of cells that have been activated in each subtype of the immune cell and overall action. Blood will also be analyzed for cortisol levels and inflammatory cytokines, (IL-1, IL-6 and TNF-alpha) using the ELISA assay procedure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, not pregnant

Exclusion Criteria:

* Fear or aversion to needles or blood draws.
* Recent infection or immunocompromised.
* Allergy to cow's milk.
* Known herb allergies.
* Aversions or medical contraindications to alcohol.
* Medication contra-indications, such as: benzodiazepines, CNS depressants,immunosuppressants and thyroid hormone and supplements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-05; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study will be to measure immune cell activation, inflammatory cytokines and cortisol levels after administration of the herb. | 24 hours and again at 5 days

SECONDARY OUTCOMES:
The secondary endpoint of this study will be to measure and correlate stress levels to the use of the herb. | 24 hours and again at 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Heather Zwickey, PhD, Principal Investigator — Helfgott Research Institute at NCNM
Locations (1):
- Helfgott Research Institute, Portland, Oregon, United States